CLINICAL TRIAL: NCT04466345
Title: Adjunctive Semaglutide for the Treatment of Cognitive Dysfunction in Major Depressive Disorder: a Randomized, Double-Blind, Placebo-Controlled Study
Brief Title: Semaglutide for the Treatment of Cognitive Dysfunction in Major Depressive Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 19-6283
Record Dates: First submitted 2020-06-08; First posted 2020-07-10 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2024-08

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Semaglutide (Experimental): Participants receive semaglutide once daily orally, initiated at 3 mg/day for 4 weeks, increased to 7 mg/day for 4 more weeks and titrated to 14 mg/day for the subsequent 8 weeks (i.e., duration of 16 weeks in total).
  Interventions: Biological: Semaglutide
- Placebo (Placebo Comparator): Participants receive matching semaglutide placebo capsules once daily (duration of 16 weeks).
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Semaglutide — 3 mg/day for 4 weeks, increased to 7 mg/day for 4 more weeks and titrated to 14 mg/day for the subsequent 8 weeks
  Arms: Semaglutide
Biological: Placebo — Semaglutide placebo capsules
  Arms: Placebo

SUMMARY:
This study will examine whether semaglutide may improve cognitive function in individuals with major depressive disorder (MDD).

DETAILED DESCRIPTION:
This is a 16-week, placebo-controlled, randomized, double-blind, clinical trial, involving 60 overweight individuals with MDD and pre-treatment cognitive dysfunction. Study participants will receive one of the following study interventions in addition to 'standard of care' treatment: once-daily semaglutide, initiated at 3 mg/day for 4 weeks, increased to 7 mg/day for 4 more weeks and titrated to 14 mg/day for the subsequent 8 weeks; or matching placebo. Participants will be assessed to examine the effect of semaglutide on their cognitive function.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent before study-related activity
2. Individuals between the ages of 18 and 60 who meet Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) criteria for MDD
3. Overweight (i.e. BMI ≥ 25 kg/m2)
4. Below-average (i.e. >1 SD below norm) performance in the Trail Making Test-B (TMTB)

Exclusion Criteria:

1. Current, or in the past 4 weeks, treatment with other oral hypoglycemic agents and/or insulin
2. Diagnosis of possible or probable Alzheimer's Disease, Mild Cognitive Impairment, or any other dementia
3. History of neurological disorder, or evidence of neurologic or other physical illness that could produce cognitive deterioration
4. Severe mood episode, defined as a Hamilton Depression Rating Scale (HAMD-17) score of >23
5. Actively suicidal or evaluated as being a suicide risk (operationalized as a score of ≥3 on HAMD-17 suicide item and/or by clinical assessment).
6. Substance use disorder within 3 months before screening or a positive baseline toxicology screen
7. DSM-5 diagnosis of obsessive compulsive disorder, posttraumatic stress disorder (current or within the last year), or borderline personality disorder as assessed by a study investigator
8. Presence of absolute or relative contraindication to semaglutide (e.g. hypersensitivity to semaglutide, hepatic impairment, renal impairment with chronic kidney disease stage 3 and above, personal or familial history of medullary thyroid cancer or Multiple Endocrine Neoplasia syndrome type 2)
9. History of diabetic retinopathy
10. History of pancreatitis or pancreatic cancer
11. Presence of clinically unstable general medical illness
12. Pregnancy or breastfeeding women

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2021-10-06 (Actual); Primary Completion 2024-12-27 (Actual); Study Completion 2024-12-27 (Actual)

PRIMARY OUTCOMES:
Executive Function Composite Score | 16 Weeks
  The primary outcome will be an executive function composite score. This score will be comprised of the Digit Symbol Substitution Test (DSST - number of symbols), the Stroop test (time to completion in the congruent and incongruent conditions), and the Spatial n-back (reaction times and accuracy in four conditions,1-back, 2-back, 3-back, and 4-back).

SECONDARY OUTCOMES:
Digit Symbol Substitution Test (DSST) | 16 Weeks
  DSST is a neurocognitive test designed to assess motor speed and concentration.
Rey Auditory Verbal Learning Test (RAVLT) | 16 Weeks
  RAVLT is a neurocognitive test designed to assess verbal learning and memory.
Stroop Test | 16 Weeks
  The Stroop Test is a neurocognitive test designed to assess the ability to inhibit cognitive interference.
Trail Making Test A (TMTA) | 16 Weeks
  TMTA is a neurocognitive test designed to assess visual scanning and attention.
Perceived Deficits Questionnaire (PDQ) | 16 Weeks
  PDQ is used to assess subjective cognitive dysfunction.
36-Item Short Form Health Survey (SF-36) | 16 Weeks
  SF-36 is used to assess quality of life.
Sheehan Disability Scale (SDS) | 12 Weeks
  SDS is used to assess functional impairment in work/school, social life, and family life.
Endicott Workplace Productivity Scale (EWPS) | 16 Weeks
  EWPS is used to assess workplace productivity.
Height | 16 Weeks
  Unit: cm
Weight | 16 Weeks
  Unit: kg
fasting glucose - Blood laboratorial marker | 16 Weeks
Diet History Questionnaire III (DHQ) | 16 Weeks
  DHQ is a freely available questionnaire used to assess dietary intake (https://epi.grants.cancer.gov/dhq3/).
Physical Activity Questionnaire (IPAQ) | 16 Weeks
  IPAQ is used to assess physical activity.
Pittsburgh Sleep Quality Index (PSQI) | 16 Weeks
  PSQI is used to assess sleep quality.
Trail Making Test B (TMTB) | 16 Weeks
  TMTB is a neurocognitive test designed to assess attention and concentration.

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo B. Mansur, MD, PhD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No